CLINICAL TRIAL: NCT05759780
Title: A Study to Test the Potential of OCT Vibrography for Measuring Biomechanical Properties of Tissues
Brief Title: OCT Vibrography for Biomechanical Properties of Tissues
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Seok Hyun Yun, Professor of Dermatology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P000338
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-05

CONDITIONS: Cornea; Skin Diseases; Gingival Diseases
Keywords: biomechanics; cornea; skin; gingiva; optical coherence tomography; vibrography
MeSH Terms: conditions — Corneal Diseases; Skin Diseases; Gingival Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy cornea (Experimental): Optical imaging of the cornea in healthy subjects
  Interventions: Device: Optical imaging of the tissues
- Healthy skin (Experimental): Optical imaging of the skin in healthy subjects
  Interventions: Device: Optical imaging of the tissues
- Healthy gingiva (Experimental): Optical imaging of the gingiva in healthy subjects
  Interventions: Device: Optical imaging of the tissues
- Keratoconus cornea (Experimental): Optical imaging of the cornea in mild and moderate keratoconus
  Interventions: Device: Optical imaging of the tissues

INTERVENTIONS:
Device: Optical imaging of the tissues — OCT vibrography

SUMMARY:
The overall goal of this study is to develop OCT Vibrography (aka OCT elastography) as a novel tool for measuring biomechanical properties of human tissues in vivo.

DETAILED DESCRIPTION:
The overall goal of this study is to develop OCT Vibrography (aka OCT elastography) as a novel tool for measuring biomechanical properties of human tissues in vivo. The investigators aim to establish baseline data in healthy subjects, compare elastic moduli in different tissue types, and measure differences in elastic moduli between keratoconus and normal eyes. If successful, this project will provide useful, previously inaccessible elastic parameters and advance the investigators' understanding of the relationship between the bulk mechanical properties and the microstructure of the human tissue in vivo. This information can ultimately be used to improve the diagnosis and treatment of keratoconus, inflammatory skin diseases, and inflammatory gingiva diseases. More broadly, the technologies developed in this project will have relevance to other potential applications beyond the tissues in this research study.

ELIGIBILITY:
Group 1:

Inclusion criteria:

• Subjects with healthy eyes (age 18 - 75, N = 50)

Exclusion criteria:

* Subjects with history of eye diseases, and previous eye surgeries.
* Subjects with diabetes, glaucoma family history
* Subjects allergic to anesthetic eyedrop, especially proparacaine
* Subjects with severe allergy
* Subjects who have difficulty biting
* Subjects who have recurrent corneal erosion

Group 2:

Inclusion criteria:

• Subjects with healthy skin (age 18 - 75, N = 10)

Exclusion criteria:

• Subjects with open cuts/sores on the skin, skin infection, or any contagious skin condition

Group 3:

Inclusion criteria:

• Subjects with healthy gingiva (age 18 - 75, N = 10)

Exclusion criteria:

• Subjects with open cuts/sores on the gingiva, gingiva infection, or any contagious gingiva condition

Group 4:

Inclusion criteria:

• Mild or moderate keratoconus subjects (age 18 - 40, N = 20)

Exclusion criteria:

• Subjects with K-max above 60 diopters (Pentacam imaging) are excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-19 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Number of subjects to successfully complete OCT Vibrography without serious unanticipated adverse events related to application of the device. | 1 year
  Frequency and severity of all treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Hyun Yun, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Background] de Sanctis U, Loiacono C, Richiardi L, Turco D, Mutani B, Grignolo FM. Sensitivity and specificity of posterior corneal elevation measured by Pentacam in discriminating keratoconus/subclinical keratoconus. Ophthalmology. 2008 Sep;115(9):1534-9. doi: 10.1016/j.ophtha.2008.02.020. Epub 2008 Apr 11. PMID 18405974
- [Background] Li X, Rabinowitz YS, Rasheed K, Yang H. Longitudinal study of the normal eyes in unilateral keratoconus patients. Ophthalmology. 2004 Mar;111(3):440-6. doi: 10.1016/j.ophtha.2003.06.020. PMID 15019316